CLINICAL TRIAL: NCT02472665
Title: Evaluation of the Pharmacokinetic Profile, Clinical Efficacy and Safety of the Von Willebrand Factor Contained in FANHDI® (Double-inactivated Human Anti-hemophilic Factor) in Pediatric Subjects With Severe Von Willebrand Disease
Brief Title: Efficacy and Safety of Fanhdi®, a High-purity Von Willebrand Containing FVIII Concentrate, in Pediatric Patients With Von Willebrand Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Collaborators: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG1005
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Von Willebrand Disease
Keywords: pediatric; plasma-derived FVIII concentrate
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- plasma-derived FVIII/VWF concentrate (Experimental): Pharmacokinetic single dose study with Fanhdi (high-purity Von Willebrand containing FVIII concentrate)
  Interventions: Drug: plasma-derived FVIII/VWF concentrate

INTERVENTIONS:
Drug: plasma-derived FVIII/VWF concentrate — 1 single dose of 80 IU/kg VWF:RCo of Fanhdi will be administered
  Other Names: Fanhdi

SUMMARY:
Multicenter, prospective, non-controlled study in a pediatric cohort (<6 years-old) with severe (type 2 or 3) hereditary Von Willebrand Disease (VWD).

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, and single-arm study. The study population is planned to include 8 pediatric subjects (<6 years of age) with severe (type 2 or 3) hereditary VWD without inhibitors and with no active bleeding at the time of inclusion. Eligible subjects will receive a single dose of Fanhdi for a PK evaluation and will be followed for 12 months for which the efficacy and safety of Fanhdi will be assessed. In addition, the type 3 VWD subjects, after 6 months of follow-up of the first infusion, will receive the second dose as in the 1st PK evaluation and undergo a 2nd PK evaluation.

The study will consist of 2 phases:

* PK profile evaluation in which all eligible subjects will receive a single dose of 80 IU/kg von Willebrand factor: Ristocetin cofactor activity (VWF:RCo) of Fanhdi. In addition, after 6 months of follow-up of the first infusion, type 3 VWD subjects will receive the second dose of Fanhdi and undergo a 2nd PK evaluation with a reduced sampling schedule.
* A 12-month Follow-up period during which the safety and efficacy of Fanhdi will be assessed in the prevention and management of bleeding episodes and/or management of perioperative hemostasis during surgery and/or invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with severe (type 2 or 3) hereditary VWD (VWF:RCo<15-20 IU/dL), or VWF:Act<15-20 IU/dL.
2. Subjects under 6 years of age.
3. Signed informed consent form (ICF) provided by an authorized representative on behalf of the subject in accordance with local law and institutional policy.

Exclusion Criteria:

1. Subjects diagnosed with acquired VWD.
2. Subjects with active bleeding at the time of the first infusion or within 10 days prior to the infusion.
3. Subjects who have been treated with DDAVP or another FVIII containing VWF concentrate during the 5 days prior to the infusion of the Fanhdi. This treatment-free period may be reduced to 3 days for subjects with type 3 VWD.
4. Subject who are positive for anti-VWF or anti-FVIII antibodies (≥0.5 Bethesda Units) or has been positive in the history of their disease.
5. Subjects with a known allergies/intolerance to any substance contained in Fanhdi.
6. Subjects with a known history of anaphylactic reaction(s) to blood or blood components.
7. Subjects presenting severe platelet activity dysfunction due to the use of drugs (aspirin, other nonsteroidal anti-inflammatory drugs [NSAIDs], etc.) or a congenital or acquired platelet function disorder or other concomitant processes that may interfere with coagulation.
8. Subjects have a known previous infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV), or have clinical signs and symptoms consistent with current HAV, HBV, HCV or HIV infection.
9. Subjects presenting anemia (hemoglobin <11 g/dL).
10. Subjects diagnosed with metabolic diseases that are not clinically controlled, such as diabetes mellitus, which could potentially interfere with the interpretations of the study.
11. Participated in another clinical trial within 30 days prior to the screening visit or has received any investigational product (IP) within 3 months prior to the screening visit.
12. If it is anticipated that the subject will be treated with other products containing FVIII or VWF different from Fanhdi throughout the subject's participation.
13. Subjects who, in the opinion of the investigator, may have compliance problems with the protocol.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
AUC^0-inf of coagulation factor VIII activity (FVIII:C) | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve extrapolated to infinity of FVIII:C
AUC^0-inf of von Willebrand factor: Ristocetin cofactor activity (VWF:RCo) | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve extrapolated to infinity of VWF:RCo
AUC^0-inf of von Willebrand factor antigen (VWF:Ag) | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve extrapolated to infinity of VWF:Ag
AUC^0-inf of von Willebrand factor: Collagen binding activity (VWF:CB) | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve extrapolated to infinity of VWF:CB
AUC^0-T of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration of FVIII:C
AUC^0-T of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration of VWF:RCo
AUC^0-T of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration of VWF:Ag
AUC^0-T of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration of VWF:CB
in vivo recovery of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
in vivo recovery of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
in vivo recovery of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
in vivo recovery of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
Half-life of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
  Terminal elimination half-life
Half-life of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
  Terminal elimination half-life
Half-life of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
  Terminal elimination half-life
C^max of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
  Maximum observed plasma and/or serum concentration of FVIII:C
C^max of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
  Maximum observed plasma and/or serum concentration of VWF:RCo
C^max of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
  Maximum observed plasma and/or serum concentration of VWF:Ag
C^max of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
  Maximum observed plasma and/or serum concentration of VWF:CB
T^max of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
  Time of maximum observed plasma and/or serum concentration of FVIII:C
T^max of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
  Time of maximum observed plasma and/or serum concentration of VWF:RCo
T^max of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
  Time of maximum observed plasma and/or serum concentration of VWF:Ag
T^max of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
  Time of maximum observed plasma and/or serum concentration of VWF:CB
Mean residence time of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
  Average amount of time that a single molecule of drug stays in the body.
Mean residence time of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
  Average amount of time that a single molecule of drug stays in the body of VWF:RCo
Mean residence time of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
  Average amount of time that a single molecule of drug stays in the body of VWF:Ag
Mean residence time of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
  Average amount of time that a single molecule of drug stays in the body of VWF:CB
Clearance of FVIII:C | Prior to the first infusion, 30 minutes postinfusion, 10 hours postinfusion, and at 24, 48, and 72 hours postinfusion
  Total plasma and/or serum clearance
Clearance of VWF:RCo | Prior to the first infusion, 30 minutes postinfusion, 10 hours postinfusion, and at 24, 48, and 72 hours postinfusion
  Total plasma and/or serum clearance
Clearance of VWF:Ag | Prior to the first infusion, 30 minutes postinfusion, 10 hours postinfusion, and at 24, 48, and 72 hours postinfusion
  Total plasma and/or serum clearance
Clearance of VWF:CB | Prior to the first infusion, 30 minutes postinfusion, 10 hours postinfusion, and at 24, 48, and 72 hours postinfusion
  Total plasma and/or serum clearance
Elimination rate constant of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
Elimination rate constant of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
Elimination rate constant of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
Elimination rate constant of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
Volume of distribution of FVIII:C | Prior to the first infusion up to 72 hours postinfusion
Volume of distribution of VWF:RCo | Prior to the first infusion up to 72 hours postinfusion
Volume of distribution of VWF:Ag | Prior to the first infusion up to 72 hours postinfusion
Volume of distribution of VWF:CB | Prior to the first infusion up to 72 hours postinfusion
VWF multimeric pattern | Prior to the first infusion up to 12 hours postinfusion
  For type 3 VWD subjects

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Sant Joan de Déu Barcelona, Esplugues de Llobregat, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided